CLINICAL TRIAL: NCT05442866
Title: Virtual Reality for Outpatient Cancer Pain Management: a Dosing Study
Brief Title: Virtual Reality for Outpatient Cancer Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004928; U2CNR014637 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Cancer Pain
MeSH Terms: conditions — Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Virtual reality (VR) dosing arm (Experimental): All participants will proceed in this single arm, in which each participant will complete baseline measures, then receive 1 week of VR daily for 10 minutes per session, then 1 week of VR twice a day for 10 minutes per session, then 1 week of VR use as desired by the participant.
  Interventions: Device: Virtual reality experience for 10 minutes

INTERVENTIONS:
Device: Virtual reality experience for 10 minutes — Each 10-minute VR session will be self-administered (by each participant) using the Facebook (Facebook Inc., Menlo Park, CA) Meta Quest 2 VR and Touch controllers. This equipment was selected because it is portable, has built in audio, and has clear graphics at a lower price than VR setups that require a computer to generate graphics. The headset has an optional eyeglass spacer to allow participants to wear corrective eyeglasses during the VR session if appropriate. The hand controllers facilitate immersive, interactive VR experiences. The VR software, Nature Treks VR application (https://naturetreksvr.com) that features ten non-violent, nature-based experiences in peaceful environments (e.g. forest, river, beach, etc.) that can be played in a seated or fixed position.

SUMMARY:
This is a non-randomized, unblinded dose-titration study to evaluate different "doses" of virtual reality to impact moderate-to-severe pain in patients living with cancer. After consenting to participate, in addition to usual pharmacologic pain management, participants will receive 1 week of VR daily for 10 minutes per session, then 1 week of VR twice a day for 10 minutes per session, then 1 week of VR use as desired by the participants.

DETAILED DESCRIPTION:
The purpose of this a non-randomized, unblinded dose-titration study to evaluate the impact of virtual reality therapy on mitigating moderate to severe pain in outpatients living with cancer.

Outpatients receiving cancer care at the Washington Cancer Institute (Washington, DC) will be considered for enrollment in this study if able to provide consent, at least 18 years old, and report moderate-severe pain (at least 4 out of 10 where pain is rated on a Likert scale between zero and 10) in the previous 7 days as a result of either cancer or cancer treatment. Palliative care consultation and/or referral to palliative care is not required for eligibility or participation. Additionally, participation will not be limited by whether subjects are receiving specific cancer-directed therapies at the time of enrollment. Subjects will be excluded if they already use VR for personal use, have intractable nausea/vomiting, history of motion sickness, history of seizures or epilepsy, have cranial structure abnormalities that prevent use of VR headset, or are currently enrolled in a palliative care or pain management study. Subjects will also be excluded if they have limited vision or vision defects that are not corrected with prescription eyeglasses, or if participants are unable or do not wish to wear required corrective eyeglasses with the VR headset. Informed consent will be conducted before enrolling each patient.

This is a non-randomized, unblinded dose-titration study. After consenting to participate, in addition to usual pharmacologic pain management, participants will receive 1 week of VR daily for 10 minutes per session, then 1 week of VR twice a day for 10 minutes per session, then 1 week of VR use as desired by the participants.

Because of the nature of the compared interventions, subjects and researchers cannot be blinded to intervention. Our primary outcome measure will determine the impact of VR on self-reported pain score in the last week (numeric rating scale, collected weekly). Self-reported pain experience remains the standard for clinical pain research. Secondary outcomes will measure pain interference (PROMIS Pain Interference Short Form, collected weekly), as-needed opioid use for patients taking opioid analgesics at the time of enrollment (self-reported using medication administration form), satisfaction with VR intervention and overall pain management (collected weekly), and survey of preferences for VR thematic content (collected after Week 4).

Following consent, subjects will complete baseline outcome assessments including self-reported pain score in the last week, the PROMIS Pain Interference Short Form, as-needed opioid use in the last week if applicable, and satisfaction with overall pain management. Subjects will then be provided with a VR headset and paired Touch controllers to bring home for the duration of the study and instructions on the frequency of use for each week. A member of the research will educate the patient on the technology and assure comfort with use. The research study coordinator will contact patients by phone at the end of each week to confirm dates and duration of use as specified by the study protocol, collect self-reported pain score in the last week, the PROMIS Pain Interference Short Form, as-needed opioid use in the last week if applicable, and satisfaction with the VR intervention and overall pain management. Additionally, participants will be surveyed on preferences for VR thematic content at the end of Week 3.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Have diagnosis of cancer (any type)
* Report moderate-severe pain related to cancer or cancer treatment at baseline
* Able to provide consent

Exclusion Criteria:

* Already use VR for personal use
* Have intractable nausea/vomiting, history of motion sickness, history of seizures or epilepsy
* Have cranial structure abnormalities that prevent use of VR headset
* Currently enrolled in a palliative care or pain management study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groninger H, Violanti D, McPherson ML, Hopkins K, Carr AL, Hurtado M, Mete M. Virtual reality for outpatient management of cancer pain: a pilot dosing study. Support Care Cancer. 2025 Jul 14;33(8):690. doi: 10.1007/s00520-025-09723-z. PMID 40653577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Reality (VR) Dosing Arm
Started | 33
Completed | 22
Not Completed | 11
Not completed — Death | 1
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Reality (VR) Dosing Arm
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Pain Score
Description: Participant reports average pain (Likert scale 0-10, 0=pain, 10=worst pain) over last 7 days; results report the average change in self-reported pain score per study week, from baseline (Study day 0) to each subsequent measurement (measured on Study day 7 (week 1), Study day 14 (week 2), Study day 21(week 3))
Time Frame: 3 weeks (baseline to Study day 21)
Measure: Mean (Standard Error); unit: score on a scale, measured each week
Arm/Group | Virtual Reality (VR) Dosing Arm
Number analyzed (Participants) | 33
score on a scale, measured each week | -0.3 (0.1)

2. Secondary Outcome: PROMIS Pain Interference Short Form
Description: Participant completes PROMIS measure of pain interference over last 7 days; PROMIS Pain Interference SF has 6 questions, each with possible scores 1 to 5, making a possible score range between 6 and 30 points - 30 points is the highest level of total pain interference, 6 points is the lowest level of total pain interference. These results report the average change in total Pain Interference SF score per study week, from baseline (Study day 0) to each subsequent measurement (measured on Study day 7 (week 1), Study day 14 (week 2), Study day 21(week 3))
Time Frame: 3 weeks (baseline to Study day 21)
Measure: Mean (Standard Error); unit: score on a scale, measured each week
Arm/Group | Virtual Reality (VR) Dosing Arm
Number analyzed (Participants) | 33
score on a scale, measured each week | -1.5 (0.4)

3. Secondary Outcome: Number of As-needed Opioid Doses Per Day
Description: Participant reports how many as-needed opioid doses used in last 7 days (only for participants prescribed as-needed opioids); results report average number of as-needed opioid doses per day for each study week
Time Frame: 3 weeks (baseline day 0 to Study day 21)
Population: Patients taking as needed opioids who completed all three study weeks
Measure: Mean (Standard Deviation); unit: prn doses per day
Arm/Group | Virtual Reality (VR) Dosing Arm
Number analyzed (Participants) | 16
prn doses per day
  prn doses per day after Week 1 | 1.6 (2.1)
  prn doses per day after Week 2 | 1.5 (2.0)
  prn doses per day after Week 3 | 1.6 (2.0)

4. Secondary Outcome: Satisfaction With Overall Pain Management
Description: Participant reports satisfaction with pain management over last 7 days (Likert scale, 0=very unsatisfied, 10=highly satisfied); results report the average change in score of overall satisfaction in pain management per study week, from baseline (Study day 0) to each subsequent measurement (measured on Study day 7 (week 1), Study day 14 (week 2), Study day 21(week 3))
Time Frame: 3 weeks (baseline to Study day 21)
Measure: Mean (Standard Error); unit: score on a scale, measured each week
Arm/Group | Virtual Reality (VR) Dosing Arm
Number analyzed (Participants) | 33
score on a scale, measured each week | 0.7 (0.2)

5. Secondary Outcome: Satisfaction With Virtual Reality Intervention Over Previous 7 Days
Description: Participant reports satisfaction with virtual reality intervention over last 7 days (Likert scale, 0=very unsatisfied, 10=highly satisfied)
Time Frame: 3 weeks (baseline to Study day 21)
Population: Patients who completed all three weeks of study completed this survey question
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Virtual Reality (VR) Dosing Arm
Number analyzed (Participants) | 22
score on a scale | 9.5 (2)

6. Secondary Outcome: Preferences for Virtual Reality Thematic Content (Measured Once, With no Comparison)
Description: Participant chooses preferred visual thematic content (as many as preferred) from photos of different images (e.g. beachscape, rain forest, luxury auto, monastery, etc.)
Time Frame: Study day 21
Population: Participants who completed all three weeks of study period
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality (VR) Dosing Arm
Number analyzed (Participants) | 22
Participants
  Prefer realistic VR | 14
  Prefer simulated VR | 7
  Prefer both/mix | 1

ADVERSE EVENTS:
Time Frame: Each participant was enrolled and followed by the study coordinator for a maximum period of 3 weeks (from enrollment and baseline measures to final measure collection). Because virtual reality has never been shown to have adverse events that last longer than the duration of the virtual reality device use, this time frame was most appropriate for adverse event data collection.
Description: Adverse events were first collected by the study coordinator during usual study processes and participant follow up and were each reviewed by the PI.
Arm/Group | Virtual Reality (VR) Dosing Arm
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 2/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Reality (VR) Dosing Arm (N=33)
Hospitalized (Infections and infestations) | 1 (1) — Participant admitted to hospital for management of infection
Surgery (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient required hospitalization and surgery for management of cancer
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Reality (VR) Dosing Arm (N=33)
Headache (General disorders) | 1 (1) — Participant experienced brief general headache during VR, headache stopped after patient stopped VR
Dizziness (Nervous system disorders) | 1 (1) — Participant experienced brief dizziness while using VR, stopped after participant stopped using VR

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT05442866/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT05442866/ICF_001.pdf